CLINICAL TRIAL: NCT00863577
Title: Pharmacokinetic Study of Two Oral Bemiparin Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rovi Pharmaceuticals Laboratories (Industry)
Responsible Party: Medical Department, Medical Department
Model: Parallel | Masking: None
Other Study IDs: ROV-BEM-2008-01
Record Dates: First submitted 2009-01-27; First posted 2009-03-18 (Estimated); Last update posted 2011-03-18 (Estimated); Status verified 2011-03

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — bemiparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Oral bemiparin — Bemiparin tablets and bemiparin tablets into hard gelatine capsules

SUMMARY:
The primary pharmacokinetic analysis will be the correlation of the AUC amidolytic anti-Xa activity

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers: male or female subjects aged between 18 and 45 years
2. Body weight: 65-80 Kg
3. Not meaningful abnormalities in physical examination and in clinical history
4. Without evidence of significant organic or psychiatric illness
5. Hemogram, biochemistry and coagulation in normal values established in the reference range of the local hospital laboratory
6. Vital signs (blood pressure, heart beat rate and body temperature) and EKG within normal range
7. Healthy volunteers who are not participating in another clinical trial or have not done so in the past 2 months
8. Not give blood in the last 4 weeks.
9. Healthy male volunteers who have not received heparin in the past
10. Healthy male volunteers who have accepted to participate in the study and have signed the written informed consent
11. contraceptive methods double barrel or sterile surgery

Exclusion Criteria:

1. Previous history of alcoholism, drug dependency, drug abuse or habitual psychoactive drugs consumption
2. Important consumption of exciting drinks: alcohol consumption > 30 g/day; coffee, tea, cola > 5 /day
3. Allergy, idiosyncrasy or hypersensitivity to medicines
4. Healthy volunteers who are receiving another medication in the past 15 days
5. Positive serology of hepatitis B, C or HIV
6. Cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, hematologic, psychiatric, neurological and others events
7. Mayor Surgery in the last 6 months
8. Smoking > 10 cigarettes / day
9. Ethanol, cannabis, cocaine, amphetamine, benzodiazepin or opiate in urine
10. Healthy volunteers with a familiar history evident hemorrhagic episodes
11. positive fecatest and comburtest
12. positive pregnant test
13. Bemiparin contraindication

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary pharmacokinetic analysis will be the correlation of the AUC amidolytic anti-Xa activity | pre-medication, +1 h , +2 h, +3h, +4 h , +5h, +6 h, +8 h, +10h, +12h, +18 h, +24 h,+25h, +26h, +27h, +28h, +29h, +30h, +32h, +34h, +36h, +42h, +48 h, +60 h and +72 h

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Santa Creu i Sant Pau, Barcelona, Barcelona, Spain